CLINICAL TRIAL: NCT03524131
Title: Randomized Controlled Trial to Compare the Effect of Two New Behaviourally Enhanced NHS Health Check Leaflets and the Current Nationally Recommended Leaflet on Uptake of NHS Health Checks
Brief Title: Randomized Controlled Trial on Uptake of NHS Health Checks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NHSHC2017
Record Dates: First submitted 2018-04-26; First posted 2018-05-14 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2018-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- risk-framed leaflet (Experimental): Patients sent 2-sided risk-framed leaflet with NHS Health Check invitation
  Interventions: Other: risk-framed leaflet
- benefits-framed leaflet (Experimental): Patients sent 2-sided benefits-framed leaflet with NHS Health Check invitation
  Interventions: Other: benefits-framed leaflet
- control (Active Comparator): Patients sent 4-sided current national leaflet with NHS Health Check invitation
  Interventions: Other: current national leaflet

INTERVENTIONS:
Other: risk-framed leaflet — 2-sided leaflet, emphasizing health risks of not going to the NHS Health Check
  Arms: risk-framed leaflet
Other: benefits-framed leaflet — 2-sided leaflet, emphasizing benefits of attending an NHS Health Check
  Arms: benefits-framed leaflet
Other: current national leaflet — 4-sided leaflet
  Arms: control

SUMMARY:
The National Health Service (NHS) Health Check is a significant part of the strategy to tackle premature mortality and promote healthy lifestyles. Public Health England aspires to an uptake rate of 75% but national uptake is less than 50%. This study aims to assess the impact of two new behaviourally informed NHS Health Check leaflets on the uptake of NHS Health Checks, by randomizing patients in Lewisham and North East Lincolnshire to the different leaflets and comparing patient-level uptake data. The study will test whether a shorter risk-framed leaflet or a shorter benefits-framed leaflet will be more effective than the current national leaflet at encouraging uptake of the NHS Health Check.

ELIGIBILITY:
Inclusion Criteria:

* due to be invited for an NHS Health Check
* aged 40-74

Exclusion Criteria:

* have an existing Cardio-Vascular Disease-related medical condition
* have had an NHS Health Check in the last five years

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
attendance at NHS Health Check | up to 6 months from time of invitation
  whether or not the patient attended their NHS Health Check

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health England, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gold N, Durlik C, Sanders JG, Thompson K, Chadborn T. Applying behavioural science to increase uptake of the NHS Health Check: a randomised controlled trial of gain- and loss-framed messaging in the national patient information leaflet. BMC Public Health. 2019 Nov 14;19(1):1519. doi: 10.1186/s12889-019-7754-5. PMID 31727030